CLINICAL TRIAL: NCT02129816
Title: Treatment of Patients With Overactive Bladder With Bryophyllum Pinnatum Versus Solifenacinsuccinat Versus Placebo: Multicenter, Prospective, Double-blind Randomized, Placebo-controlled Cross-over Study, Phase III Trial
Brief Title: Bryophyllum Pinnatum Versus Solifenacin Versus Placebo for Overactive Bladder
Acronym: BryoSoliP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: PD Dr. med. Verena Geissbühler (Unknown); Prof. pharm. Ursula von Mandach (Unknown); Dr. med. David Scheiner (Unknown); Dr. med. Matthias Werner (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BryoSoliP-2014; KEK 2012-0530 (Zurich) (Registry Identifier: Ethics committee Zurich)
Record Dates: First submitted 2014-04-25; First posted 2014-05-02 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Overactive Bladder; Urge Urinary Incontinence
Keywords: Female; Postmenopause
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bryophyllum (Active Comparator): 50% in 350mg Lactose, 2-2-2
  Interventions: Drug: Bryophyllum
- Placebo (Placebo Comparator): Lactose 350mg, 2-2-2
  Interventions: Drug: Bryophyllum
- Solifenacin (Experimental): 10mg in 350mg Lactose, 2-2-2
  Interventions: Drug: Bryophyllum

INTERVENTIONS:
Drug: Bryophyllum
  Other Names: dried leave press juice; provided by Weleda AG, Arlesheim, Switzerland

SUMMARY:
Overactive bladder (OAB) is an enigmatic condition that is treated symptomatically with anticholinergic drugs (gold standard 2013). In a clinical pilot study was found to be a trend for a higher reduction of the micturition frequency in the Bryophyllum pinnatum group - treated with chewing tablets containing 50% of dried BP leaf press juice - than in the placebo group (n=20, p=0.064) Hypothesis: To test the superior effectivity of Bryophyllum versus Placebo in the treatment of OAB with the needed number (Purpose 1) and to assess in an experimental arm the side effects of BP in comparison to the standard drug (Vesicare) in a clincial trial (Purpose 2).

DETAILED DESCRIPTION:
* In a US nation-wide survey, lower urinary tract symptoms are one of the strongest predictors that patients will seek complementary and alternative medicine (CAM) care. In comparison to general gynecological patients, urogynecological patients are particularly prone to seek help in CAM. Moreover out of the different CAM options, herbal medication is one of the most preferred treatments. However, the effectiveness of CAM regarding OAB has not yet been adequately and objectively evaluated. Therefore, it is timely and essential to elucidate the mode of action as well as to prove efficacy of herbal treatments by a translational approach including comprehensive in vitro experimentation and randomized controlled clinical trials. Bryophyllum pinnatum and specially the flavonoid components have shown a muscle relaxing effect on porcine bladder strips.
* Study Design: Multicenter, prospective, double-blind randomized, placebo-controlled cross-over study, phase III to test the superiority of Bryophyllum pinnatum (BP) over placebo in the treatment of overactive bladder.
* In this cross-over trial a total of 30 patients is needed to proof the superiority of BP over placebo (5 randomization blocs, each 6 patients). Each patient gets each of the three study drugs (BP, Solifenacin, Placebo) in a double-blind randomization. The number of patients was calculated in a post-hoc analysis based on the primary endpoint of a previous study (reduction of micturition rates/24hours; 9.5 (SD2.2) before and 7.8 (SD1.2) after Bryophyllum versus 9.3 (SD1.8) before and 9.1(SD1.6) after placebo), under the assumption of a normal data distribution and a power of 80% a patient number of 2x20. Plus 10% for non-parametric tests in the case of a non-normal distribution (Wilcoxon) were added, what generated a number of 2x22 patients.
* In order to facilitate an equality in the randomization, the investigator choose a cross-over design. Due to the length of the study time, the drop-out rate was risen from 10 to 20% what yielded under the assumption of a equal block randomization the number of 30 patients. Additionally, an explorative arm containing the standard medication Vesicare was inserted, as this is of great clinical interest. For this explorative comparative arm are no existing data that would allow to do a power calculation.
* This follow-up study will give a compelling answer on the efficacy or non-efficacy of BP as well as the safety of BP in respect to placebo and possible answers of its position regarding the standard medication Vesicare.

ELIGIBILITY:
Inclusion Criteria:

* OAB (>8 micturitions/24 hours, associated with urge symptoms)
* postmenopausal women
* cystoscopy to exclude a bladder carcinoma or carcinoma in situ
* written and oral informed consent

Exclusion Criteria:

* urinary tract infection in an intermittent catheter asservated sample (>1000 bacterias/ml)
* intake of bladder affecting drugs like anticholinergics, diuretics, muscle relaxing medications and phytotherapeutics in the last three months
* neurological conditions such as stroke, multiple sclerosis, spinal cord injury or Parkinsons's disease
* postvoid residual volume ≥100 ml
* lactose intolerance
* contraindication for Solifenacin

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04-20 (Actual); Study Completion 2017-07-09 (Actual)

PRIMARY OUTCOMES:
Change of the micturition frequency | participants will be followed for the duration of the study, an expected average of 35 weeks
  assessment of the voiding frequency in the 3-day bladder at visit 2,3,4,5,6

SECONDARY OUTCOMES:
Changes in quality of life parameters | participants will be followed for the duration of the study, an expected average of 35 weeks
  assessment with quality of life and symptom burden questionnaires at visit 2,3,4,5,6 (questionnaires ICIQ-OAB and KHQ)
Voiding diary parameters | participants will be followed for the duration of the study, an expected average of 35 weeks
  3-day bladder diary returned at visit 2,3,4,5,6
Assessments of the patient's compliance | participants will be followed for the duration of the study, an expected average of 35 weeks
  drug intake protocol and counting of the returned tablets
Assessment of AE/SAE | participants will be followed for the duration of the study, an expected average of 35 weeks
  AE/SAE protocol

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Gynecologic Department, University Hospital Zurich, Zurich
  - Gynecology Department, University Hospital Zurich, Zurich

REFERENCES:
- [Result] Betschart C, von Mandach U, Seifert B, Scheiner D, Perucchini D, Fink D, Geissbuhler V. Randomized, double-blind placebo-controlled trial with Bryophyllum pinnatum versus placebo for the treatment of overactive bladder in postmenopausal women. Phytomedicine. 2013 Feb 15;20(3-4):351-8. doi: 10.1016/j.phymed.2012.10.007. Epub 2012 Dec 4. PMID 23218404